CLINICAL TRIAL: NCT01305967
Title: Phase Ⅱa,Open Label,Multicenter Clinical Trial to Investigate Safety and Efficacy of SB Injection in Patients With Advanced and Metastatic Non-small Cell Lung Cancer
Brief Title: Investigation of Safety and Efficacy of SB Injection in Patients With Advanced and Metastatic Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SBPharmaceutical IND, Co., LTD (Industry)
Responsible Party: Lee Dong-heum / executive director, SBPharmaceutical IND, Co., LTD
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB Injection
Record Dates: First submitted 2011-02-24; First posted 2011-03-01 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB injection — Infusion SBinjection of 21.87ml/m^2, Intravenous route, 16times for 2.5 months

SUMMARY:
The purpose of this study is to determine efficacy of SB injection in Non Small Cell Lung Cancer.

DETAILED DESCRIPTION:
All eligible patients will receive SB injection therapy for 4 cycles (14~21 days for each cycle). SB injection treatment could be continue after completion of therapy cycles until 6th cycle. It depends on the investigator's decision and patient's will. Efficacy will be evaluated every two cycles.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-70 years
* Patients with histologically or cytologically confirmed Non-Small Cell Lung Cancer
* Patients who had failed more than 1 cycle of standard therapy with advanced or metasatic stage not available to any of resectable surgery or radiotherapy.
* Patients with measurable lesions
* Eatern Cooperative Oncolgy Group status 0 to 2.
* Life expectancy >/= 5 months
* Patients with adequate organ(heart, kidney, liver)and bone marrow function, as defined by

  1. Absolute neutrophil count >/= 1.5 x 10^9/L, Platelet count >/= 100 x 10^9/L
  2. Total bilirubin </= upper limit of normal
  3. Aspartate Aminotransferase and/or Alanine Aminotransferase </= 2 x upeer limit of normal
  4. creatinine </= 1.5 x upeer limit of normal
* Patients who have signed the informed consent form.

Exclusion Criteria:

* Female volunteers admitted to the study must be using a reliable means of contraception
* Received radiation therapy within 6 weeks before randomization
* Known brain or spinal cord metastases
* Have acute infection
* Have active infection or serious concomitant systemic disorder incompatible with the study
* Presence or history of malignancy other than Non-Small Cell Lung Cancer
* Have severe neurologic or psychological disorder
* Patients who have to receive other chemo-radiotherapy or immunotherapy
* Patients who have received chemotherapy within the previous 30 days
* Patients who are candidates for combined modality treatment.
* Patients who have participated in a clinical study within the previous 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2003-01; Primary Completion 2011-05 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Overall Best Response Rate | 2.5 months

SECONDARY OUTCOMES:
Determine duration of response rate by measuring time to progression | 2.5 months
Pain Scores on the Visual Analog Scale | 2.5months
Evalute patient's performance by measuring the Eastern Cooperative Oncology Group scale | 2.5months

CONTACTS AND LOCATIONS:
Overall Officials: Jae-yong Park, Professor, Principal Investigator — Kyungpook University Hospital; Seung-beom Han, Professor, Principal Investigator — Keimyung University Dongsan Medical Center; Chae-young Lee, Medical Doctor, Principal Investigator — Anyang Sam Medical Center
Locations (3):
- South Korea (3):
  - Keimyung University Dongsan Hospital, Daegu, Jung-gu
  - Kyungpook University Hospital, Deagu, Jung-gu
  - Sam Anyang Medical Center, Anyang, Man-an-gu

REFERENCES:
- See also: SBP — http://www.sbp.com/